CLINICAL TRIAL: NCT01944826
Title: A Prospective, Multicenter, Observational Registry to Evaluate the Prevalence and Incidence of Cancer and Long-term Prognosis in Patients With Tako-Tsubo (Stress-induced) Cardiomyopathy.
Brief Title: The TAKO-TSUBO And Cancer Registry
Acronym: TTAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: TTAC
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Tako-Tsubo Cardiomyopathy; Stress-induced Cardiomyopathy; Acute Coronary Syndrome
Keywords: Dyspnea; Angina pectoris
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Acute Coronary Syndrome; Dyspnea; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Laboratory parameters and biomarkers:
  * Faecal occult blood test
  * Complete blood count including erythrocyte sedimentation rate
  * Serum protein electrophoresis
  * Prostate-specific antigen (PSA) testing in men
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tako-Tsubo And Cancer Registry
  Interventions: Other: Registry of patients with Tako-Tsubo cardiomyopathy

INTERVENTIONS:
Other: Registry of patients with Tako-Tsubo cardiomyopathy

SUMMARY:
Prospective, multicenter, observational registry collecting data from subjects with Tako-Tsubo (stress-induced) cardiomyopathy (TTC). Uniform, complete, and accurate data will be collected on the subject's medical history, during index hospitalization for TTC, and during follow-up.

The objectives are to evaluate the prevalence and incidence of cancer in patients with TTC, to document the underlying causes of death during hospital stay and during follow-up, to determine the long-term prognosis, and to identify possible predictors of short and long-term mortality.

DETAILED DESCRIPTION:
The prognosis of patients with TTC is believed to be favorable. This assumption is mainly based on the observations of a rapid recovery of global left ventricular function and low cardiac in-hospital mortality. In fact, the clinical course following TTC events after hospital discharge is largely unknown due to a lack of large prospective long-term follow-up studies and inconsistent and limited findings from available studies to date.

The TTAC registry represents the first attempt to initiate an international registry with special focus on comorbidities, particularly malignancies, in patients with TTC to further elucidate the relationship between these diseases. In addition, the TTAC registry will enable documenting the exact underlying causes of death and long-term prognosis of patients with TTC and to identify possible predictors of short and long-term mortality in these patients.

The first objective of this prospective, multicenter, observational registry is to evaluate the prevalence and incidence of cancer in patients with TTC.

The second objective is to document the underlying causes of death during hospital stay and follow-up and to determine the long-term prognosis of patients with TTC.

The third objective is to identify possible predictors of short and long-term mortality in patients with TTC.

Available information is collected from subjects being treated according to routine clinical practice. In addition, during the index hospitalization, each subject is screened for occult cancer disease. During follow-up, cancer screening will be performed according to appropriate legal preventive examinations.

Subjects will be followed at 6 months and annually after the index event for up to 5 years by phone call, office visit, or by contacts with primary physicians or referring cardiologists, according to each investigator's preference.

As regulated by data protection and privacy laws and in accordance with local ethics committee requirements, subjects will be informed and requested to grant their approval after the index procedure (= cardiac catheterization for suspected acute coronary syndrome) to review their medical records and collect and analyze personal medical information. The confidentiality of the records will be maintained at all times. Subjects will be asked to agree to perform a cancer screening during index hospitalization and will also be asked to agree to be contacted during the 5-year follow-up period.

Patients in whom TTC was diagnosed will be informed and requested to grant their approval to review their medical records, to collect and analyze personal medical information, while maintaining the confidentiality of the records at all times. Subjects will be asked to agree to perform a cancer screening during index hospitalization and will also be asked to agree to be contacted during the 5-year follow-up period. Informed consent will be requested after the index procedure (= cardiac catheterization for suspected acute coronary syndrome proving presence of TTC) and the informed consent form (ICF) has to be signed prior to entering subject's data in the database or prior to any follow-up contact, whichever occurs first.

The investigator and/or designee must clearly document the process of obtaining informed consent in the subject's source documents. The voluntary process of obtaining informed consent confirms the subject's willingness to participate in the registry. It is the investigator's responsibility to ensure that the informed consent process is performed in accordance with Good Epidemiological Practice (GEP) - IEA Guidelines for proper conduct of epidemiological research and where applicable country regulations.

Subjects will be followed at 6 months and annually after the index event for up to 5 years by phone calls, office visits, or by contacts with general practitioners or referring cardiologists, according to each investigator's preference.

ELIGIBILITY:
Inclusion Criteria:

* Tako-Tsubo (stress-induced) cardiomyopathy (TTC)

Exclusion Criteria:

* myocardial infarction/ heart attack

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be collected on approximately 800 subjects with TTC.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
prevalence and incidence of cancer in patients with TTC | 5 years

SECONDARY OUTCOMES:
causes of death during hospital stay and during follow-up | 5 years

OTHER OUTCOMES:
possible predictors of short and long-term mortality in patients with TTC | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christof Burgdorf, Dr., Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum München, Munich, Bavaria, Germany